CLINICAL TRIAL: NCT01238939
Title: A Phase I Study of NK012 in Combination With Infusional 5-fluorouracil and Leucovorin in Patients With Advanced Solid Tumors Followed by a Dose Expansion Phase in Patients With Metastatic Colorectal Cancer
Brief Title: Study of NK012 and 5-FU/LV in Solid Tumors Followed by Dose Expansion in Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6012113US
Record Dates: First submitted 2010-11-02; First posted 2010-11-11 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Advanced Solid Tumors; Metastatic Colorectal Cancer
Keywords: solid tumors; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: NK012 and 5-FU

INTERVENTIONS:
Drug: NK012 and 5-FU — NK012 infusion on Day 1 of each 28 day cycle 5-FU continuous infusion on Days 1 and 15 of each 28 day cycle

SUMMARY:
The primary objective is to determine the maximum tolerated dose/recommended phase II dose of the combination regimen of NK012 and 5-fluorouracil in patients with advanced solid tumors.

DETAILED DESCRIPTION:
On Day 1 of each 28 day cycle, NK012 will be administered as a 30 minute IV infusion, followed by continuous infusion of 5-FU over 46 hours. On Day 15 of each cycle, patients again receive 5-FU continuous infusion. Treatment is expected to continue for 6 cycles, unless disease progression or the development of unacceptable toxicity requires discontinuation of the drug. At the discretion of the investigator, patients who show signs of benefit may continue beyond 6 cycles.

Once a MTD/RD has been determined for the combination regimen, a dose expansion cohort of patients with metastatic colorectal cancer will be treated at the determined MTD.

(Prior to Amendment 2, patients were receiving NK012 and 5-FU and leucovorin (LV). The dosing regimen was changed as of Amendment 2 to NK012 and 5-FU.)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of advanced solid tumor for which no efficacious therapy exists, or for which a camptothecin-based regimen would be appropriate.
2. For the dose expansion at MTD/RD only:

   1. The patient must have failed oxaliplatin-based first line therapy for metastatic colorectal cancer. This includes patients who failed oxaliplatin-based therapy with progressive disease, as well as patients who, based on toxicity or MD/patient discretion, are no longer candidates for oxaliplatin. Patients who failed adjuvant therapy with oxaliplatin-based chemotherapy regimens within one year of last dose of oxaliplatin-based chemotherapy will also be considered eligible for this study.
   2. Patients must have had no more than one prior chemotherapy regimen in the metastatic setting. Patients who had radiosensitizing chemotherapy during radiation treatment will not have this treatment count as a prior chemotherapy regimen.
   3. Patients must have measurable disease by RECIST (version 1.1).
3. Patient must have recovered from all acute adverse effects of prior therapies, excluding alopecia.
4. For patients enrolled in the dose escalation phase, no more than 4 prior cytotoxic regimens in the metastatic setting.
5. Prior irradiation to no more than 25% of the bone marrow.
6. ECOG performance status of 0-1.
7. Life expectancy of at least 12 weeks.
8. Patients are at least 18 years of age.
9. Adequate bone marrow function as defined by ANC ≥ 1500/mm^3 and platelet count ≥ 100,000/mm^3.
10. AST and ALT ≤ 3.0 x ULN (5 x ULN if documented liver metastases) and total bilirubin ≤ 1.5 x ULN.
11. Serum creatinine ≤ 1.5 x ULN, or creatinine clearance ≥ 60 mL/min by Cockcroft-Gault formula* for patients with serum creatinine > 1.5 x ULN.

    *Cockcroft-Gault formula for creatinine clearance (CrCl): Males: CrCl (ml/min) = (140 - age) x wt (kg) / (serum creatinine x 72) Females: Multiply the above result by 0.85
12. Able to understand and show willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior chemotherapy, radiation therapy, or investigational therapy within 4 weeks (exception: 6 weeks for nitrosoureas or mitomycin C); or prior non-cytotoxic therapy within 5 drug half-lives (or 4 weeks, which ever is shorter); or monoclonal antibodies within 4 weeks prior to the first dose of study treatment.
2. Concurrent use of other investigational agent.
3. History of brain metastases or spinal cord compression, unless irradiated or treated a minimum of 4 weeks prior to first study treatment and stable without requirement of corticosteroids for > 1 week.
4. Concurrent serious infections requiring parenteral antibiotic therapy.
5. Pregnant or of childbearing potential and not using methods to avoid pregnancy. A negative pregnancy test must be documented at baseline for women of childbearing potential. Patients may not breast-feed infants while on this study.
6. Significant cardiac disease including heart failure that meets NYHA class III and IV definitions, history of myocardial infarction within 6 months of study entry, uncontrolled dysrhythmias or poorly controlled angina.
7. History of serious ventricular arrhythmia (VT or VF, ≥ 3 beats in a row), QTc ≥ 450 msec for men and 470 msec for women, or LVEF ≤ 40% by MUGA or ECHO.
8. History of allergic reactions attributed to compounds of topoisomerase I inhibitors.
9. Prior treatment with irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity as determinant of the maximum tolerated dose/recommended dose | From date of first dose to off-study (or 30 days since last dose)

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | From date of first dose to off-study (or 30 days since last dose)
Tumor measurements, as a measure of efficacy | Baseline, then every on average every 2 months until off-study
  Efficacy, based on RECIST 1.1, will be assessed in all solid tumors, and in a specific subset of patients with colorectal cancer
Area under the plasma concentration versus time curve (AUC) of NK012 and fluorouracil | 15,30min, 1,6,24,46.5,48,72hrs, Wk1,2,3,4 of cycle 1
Peak Plasma Concentration (Cmax) of NK012 and fluorouracil | 15,30min, 1,6,24,46.5,72hrs, week 1,2,3,4 of cycle 1

CONTACTS AND LOCATIONS:
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States